CLINICAL TRIAL: NCT01757288
Title: A RANDOMIZED PHASE I/II STUDY OF NAB-PACLITAXEL, OR PACLITAXEL, PLUS CARBOPLATIN WITH CONCURRENT RADIATION THERAPY FOLLoWED BY CONSOLIDATION IN PATIENTS WITH FAVORABLE PROGNOSIS INOPERABLE STAGE IIIA/B NON-SMALL CELL LUNG CANCER (NSCLC)
Brief Title: Phase I/II NabPaclitaxel, Paclitaxel&Carboplatin w RTX Followed by Consolidation in Patients w Favorable Prognosis Inoperable Stage IIIA/B NSCLC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Celgene (Industry)
Responsible Party: Principal Investigator, Yuanyuan Zhang, Instructor of Department of Radiation Oncology, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU 062012-053
Record Dates: First submitted 2012-12-20; First posted 2012-12-28 (Estimated); Results first posted 2021-10-05 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: STAGE IIIA/B NSCLC / INOPERABLE LUNG CANCER
Keywords: STAGE IIIA/B NSCLC / INOPERABLE LUNG CANCER
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — 130-nm albumin-bound paclitaxel; Paclitaxel

STUDY DESIGN:
Intervention Model Description: This is Phase I/II study. Phase I has 1 arm and Phase II has 2 arms (total 3 arms)
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PACLITAXEL (Phase II, Arm A) (Active Comparator): PACLITAXEL PLUS CARBOPLATIN WITH CONCURRENT RADIATION THERAPY
  Interventions: Drug: PACLITAXEL
- NAB-PACLITAXEL (Phase II, Arm B) (Experimental): NAB-PACLITAXEL PLUS CARBOPLATIN WITH CONCURRENT RADIATION THERAPY nab-Paclitaxel 40 mg/m2 IV/30min/wk x6 wks
  Interventions: Drug: NAB-PACLITAXEL
- NAB-PACLITAXEL (Phase I) (Experimental): NAB-PACLITAXEL PLUS CARBOPLATIN WITH CONCURRENT RADIATION THERAPY nab-Paclitaxel 50 mg/m2 IV/30min/wk x6 wks
  Interventions: Drug: NAB-PACLITAXEL

INTERVENTIONS:
Drug: NAB-PACLITAXEL — nab-Paclitaxel 50 mg/m2 IV/30min/wk x6 wks
  Other Names: Abraxan
  Arms: NAB-PACLITAXEL (Phase I)
Drug: PACLITAXEL
  Arms: PACLITAXEL (Phase II, Arm A)
Drug: NAB-PACLITAXEL — nab-Paclitaxel 40 mg/m2 IV/30min/wk x6 wks
  Other Names: Abraxan
  Arms: NAB-PACLITAXEL (Phase II, Arm B)

SUMMARY:
The investigators propose this phase I/II study to use weekly Nab-Paclitaxel (Abraxane) and carboplatin with concurrent radiation in local-regionally advanced lung cancer. There are no published human studies combining Nab-Paclitaxel (Abraxane) with radiation. The investigators will first confirm the tolerated dose (TD) of concurrent Nab-Paclitaxel (Abraxane) at 50mg/m2, and then will begin enrolling patients into the phase II component using either Nab-Paclitaxel (Abraxane) at the TD with carboplatin concurrent with daily radiation or paclitaxel with carboplatin concurrent with daily radiation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented NSCLC; Patients must be M0. Patients with T1-T2 with N2 or T3N1-2 are eligible, if inoperable. Patients with T4 with any N or any T with N2 or N3 disease are eligible if unresectable.
* Patients with tumors adjacent to a vertebral body are eligible as long as all gross disease can be encompassed in the radiation boost field. The boost volume must be limited to < 50% of the ipsilateral lung volume.
* Patients with Zubrod performance status 0-1
* Adequate hematologic function
* FEV1 with ≥ 1200 cc or ≥ 50% predicted

Exclusion Criteria:

* Prior systemic chemotherapy (for lung cancer) and/or thoracic/neck radiotherapy for any reason and/or surgical resection of present cancer
* Exudative, bloody, or cytologically malignant effusions
* Prior therapy with any molecular targeted drugs (for lung cancer)
* Active pulmonary infection not responsive to conventional antibiotics
* Clinically significant cardiovascular event (e.g. myocardial infarction, superior vena cava syndrome (SVC), New York Heart Association (NYHA) classification of heart disease >2 (see Appendix B) within 3 months before entry; or presence of cardiac disease that, in the opinion of the Investigator, increases the risk of ventricular arrhythmia.
* Patients with > grade 1 neuropathy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2013-03-25 (Actual); Primary Completion 2019-06-03 (Actual); Study Completion 2019-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuanyuan Zhang, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (5):
- United States (5):
  - University of Rochester, Rochester, New York
  - UPMC Cancer Center, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 6 patients enrolled in phase I and 92 patients enrolled in phase II, 46 patints were randomized to Arm A, and 46 patients to Arm B.
Groups:
- NAB-PACLITAXEL (Phase I): NAB-PACLITAXEL PLUS CARBOPLATIN WITH CONCURRENT RADIATION THERAPY nab-Paclitaxel 50 mg/m2 IV/30min/wk x6 wks
  Carboplatin AUC **2 IV/30 min/wk x6wks XRT 6000 cGy
- PACLITAXEL (Phase II, Arm A): PACLITAXEL PLUS CARBOPLATIN WITH CONCURRENT RADIATION THERAPY Paclitaxel 50 mg/m2 IV/1h/wk* x6 wks Carboplatin AUC **2 IV/30 min/wk x6 wks XRT 6000 cGy
- NAB-PACLITAXEL (Phase II, Arm B): NAB-PACLITAXEL PLUS CARBOPLATIN WITH CONCURRENT RADIATION THERAPY nab-Paclitaxel 40 mg/m2 IV/30min/wk x6 wks Carboplatin AUC **2 IV/30 min/wk x6 wks XRT 6000 cGy
Period: Overall Study
Arm/Group | NAB-PACLITAXEL (Phase I) | PACLITAXEL (Phase II, Arm A) | NAB-PACLITAXEL (Phase II, Arm B)
Started | 6 | 46 | 46
Completed | 6 | 38 | 37
Not Completed | 0 | 8 | 9
Not completed — Consent withdrawal | 0 | 4 | 4
Not completed — Patient off study, IRB hold. | 0 | 0 | 1
Not completed — Patient death prior to starting treatment | 0 | 0 | 1
Not completed — Wrong medication administered | 0 | 1 | 0
Not completed — Liver metastasis identified at CT simulation | 0 | 1 | 0
Not completed — Not meeting protocol constraints | 0 | 1 | 1
Not completed — Multiple missed appointments | 0 | 1 | 0
Not completed — Mulitple hospitalization ( after first week of CRT) | 0 | 0 | 1
Not completed — >2 weeks treatment break | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: 75 patients were eligible for analysis on the phase II portion
Groups:
- Total: Total of all reporting groups
Arm/Group | NAB-PACLITAXEL (Phase I) | PACLITAXEL (Phase II, Arm A) | NAB-PACLITAXEL (Phase II, Arm B) | Total
Number analyzed (Participants) | 6 | 46 | 46 | 98
Age, Customized [Median (Full Range); unit: months,years]
  Median age, years | 64 [59 to 77] | 65.5 [41 to 87] | 66.5 [44 to 86] | 66 [41 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 26 | 20 | 48
  Male | 4 | 20 | 26 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 6 | 45 | 45 | 96
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 0 | 3 | 6 | 9
  White | 6 | 41 | 38 | 85
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: 2-year Overall Survival (Phase II)
Description: 2-year overall survival, as measured (by Kaplan-Meir method) as the percentage of patients who were randomized and received carboplatin/paclitaxel or carboplatin/nab-paclitaxel with radiation therapy survived for 2 years.
Time Frame: 2 years
Population: This outcome was collected for Phase II participants only 2- year overall survival.
Measure: Mean (Full Range); unit: percentage of participants
Arm/Group | NAB-PACLITAXEL (Phase I) | PACLITAXEL (Phase II, Arm A) | NAB-PACLITAXEL (Phase II, Arm B)
Number analyzed (Participants) | 0 | 38 | 37
percentage of participants |  | 66.5 [48.4 to 79.5] | 55.5 [36.3 to 71.0]

2. Secondary Outcome: The Feasibility of Concurrent Carboplatin/Nab-Paclitaxel and Radiation Therapy
Description: The feasibility as measured by the number of participants who had grade 3 or higher radiation related esophagitis or pulmonary toxicity or chemotherapy related grade 4 hematological or other non-hematological toxicities occurring within 60 days of the start of treatment; compliance us defined as the completion of the treatment regimen with no more than minor variations.
Time Frame: 60 days of the start of treatment
Population: This outcome was collected for Phase I participants only. (6 total).
Measure: Count of Participants; unit: Participants
Arm/Group | NAB-PACLITAXEL (Phase I) | PACLITAXEL (Phase II, Arm A) | NAB-PACLITAXEL (Phase II, Arm B)
Number analyzed (Participants) | 6 | 0 | 0
Participants | 0 |  |

3. Secondary Outcome: Overall Response Rate for the Patients Receiving Carboplatin/ Paclitaxel or Carboplatin/ Nab-paclitaxel With Radiation Therapy
Description: The objective response rate (ORR) is defined as the percentage of participants achieving complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST1.1) criteria
Time Frame: 1,6,12,18,24 month
Population: This outcome was measured from Phase II participants only. Percent CR/PR rates by treatment arm.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NAB-PACLITAXEL (Phase I) | PACLITAXEL (Phase II, Arm A) | NAB-PACLITAXEL (Phase II, Arm B)
Number analyzed (Participants) | 0 | 38 | 37
percentage of participants
  1 month scan |  | 36.8 [21.8 to 54.0] | 45.9 [29.5 to 63.1]
  6 month scan |  | 21.1 [9.6 to 37.3] | 24.3 [11.8 to 41.2]
  12 month scan |  | 10.5 [2.9 to 24.8] | 13.5 [4.5 to 28.8]
  18 month scan |  | 10.5 [2.9 to 24.8] | 5.4 [0.7 to 18.2]
  24 month scan |  | 2.6 [0.1 to 13.8] | 8.1 [1.7 to 21.9]

4. Secondary Outcome: Proportion of Participants With Progression-free Survival (Phase II)
Description: Proportion of participants with progression free survival at 2 years is computed as the percentage of participants between randomization and local or regional progression, distant metastases, death, or last known follow-up. Estimates of progression free survival will be calculated using the Kaplan-Meir method.
Time Frame: 2 years
Population: This outcome was collected from Phase II participants only
Measure: Median (Full Range); unit: percentage of participants
Arm/Group | NAB-PACLITAXEL (Phase I) | PACLITAXEL (Phase II, Arm A) | NAB-PACLITAXEL (Phase II, Arm B)
Number analyzed (Participants) | 0 | 38 | 37
percentage of participants |  | 44.4 [27.6 to 59.9] | 27.3 [13.7 to 42.9]

5. Secondary Outcome: Median Overall Survival (Phase II)
Description: Median overall survival was based on the Kaplan-Meier method is defined as the time from study entry to death or censored at date last known alive.
Time Frame: every 6 months up to 24 months (approx. 22 months)
Population: This outcome was measured from Phase II participants only.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | NAB-PACLITAXEL (Phase I) | PACLITAXEL (Phase II, Arm A) | NAB-PACLITAXEL (Phase II, Arm B)
Number analyzed (Participants) | 0 | 38 | 37
months |  | NA [0 to 0] — Median survival rate not reached by any of the participants enrolled in this arm | 27.8 [16.8 to 37.8]

6. Secondary Outcome: EuroQol-5Dimension (EQ-5D) MUS Score at Baseline
Description: EQ-5D is a two-part questionnaire. The first part of mean utility score (MUS) consists of five items addressing five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension can be graded on three levels: 1-no problems, 2- slight problems, and 3-moderate problems, 4-severe problems, 5-extreme problems.
  Possible score ranges from 5-25 with higher scores indicating worse outcome.Both the five-item index score and the VAS score are transformed into a utility score between 0-"worst health state" and 1-"best health state."
Time Frame: Baseline
Population: This outcome was measure from Phase II participants only
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | NAB-PACLITAXEL (Phase I) | PACLITAXEL (Phase II, Arm A) | NAB-PACLITAXEL (Phase II, Arm B)
Number analyzed (Participants) | 0 | 38 | 37
score on a scale |  | 0.49 [0.40 to 0.57] | 0.44 [0.39 to 0.50]

7. Secondary Outcome: EuroQol-5Dimension (EQ-5D) MUS Score at End of Treatment
Description: EQ-5D is a two-part questionnaire. The first part of mean utility score (MUS) consists of five items addressing five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension can be graded on three levels: 1-no problems, 2- slight problems, and 3-moderate problems, 4-severe problems, 5-extreme problems.
  Possible score ranges from 5-25 with higher scores indicating worse outcome. Both the five-item index score and the VAS score are transformed into a utility score between 0-"worst health state" and 1-"best health state."
Time Frame: End of treatment (6 weeks)
Population: This outcome was measure from Phase II participants only
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | NAB-PACLITAXEL (Phase I) | PACLITAXEL (Phase II, Arm A) | NAB-PACLITAXEL (Phase II, Arm B)
Number analyzed (Participants) | 0 | 38 | 37
score on a scale |  | 0.55 [0.44 to 0.67] | 0.45 [0.39 to 0.52]

8. Secondary Outcome: EuroQol-5Dimension (EQ-5D) VAS Score at Baseline
Description: The second part of the EQ-5D is a visual analogue scale (VAS) valuing current health state, measured on a 20-cm 10-point-interval scale.
  Worst imaginable health state is scored as 0 at the bottom of the scale, and best imaginable health state is scored as 100 at the top.
  Possible score ranges from 0-100 with higher scores indicating better outcome.
Time Frame: Baseline
Population: This outcome was measure from Phase II participants only
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | NAB-PACLITAXEL (Phase I) | PACLITAXEL (Phase II, Arm A) | NAB-PACLITAXEL (Phase II, Arm B)
Number analyzed (Participants) | 0 | 38 | 37
score on a scale |  | 0.80 [0.72 to 0.88] | 0.79 [0.72 to 0.87]

9. Secondary Outcome: EuroQol-5Dimension (EQ-5D) VAS Score at End of Treatment
Description: as for outcome 8
Time Frame: End of Treatment (6 weeks)
Population: This outcome was measure from Phase II participants only
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | NAB-PACLITAXEL (Phase I) | PACLITAXEL (Phase II, Arm A) | NAB-PACLITAXEL (Phase II, Arm B)
Number analyzed (Participants) | 0 | 38 | 37
score on a scale |  | 0.64 [0.50 to 0.79] | 0.78 [0.71 to 0.86]

10. Secondary Outcome: EuroQol-5Dimension (EQ-5D) VAS Score at 24 Month Follow up
Description: as for outcome 8
Time Frame: 24 month follow up
Population: This outcome measure was only collected for one participant a 24 months due to all other participants not completing the QOL timepoint
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | NAB-PACLITAXEL (Phase I) | PACLITAXEL (Phase II, Arm A) | NAB-PACLITAXEL (Phase II, Arm B)
Number analyzed (Participants) | 0 | 1 | 0
score on a scale |  | 0.6 [0.6 to 0.6] |

11. Secondary Outcome: EuroQol-5Dimension (EQ-5D) MUS Score at 24 Month
Description: as for outcome 6
Time Frame: 24 month follow up
Population: This outcome measure was only collected for one participant a 24 months due t oall other participants not completing the QOL timepoint
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | NAB-PACLITAXEL (Phase I) | PACLITAXEL (Phase II, Arm A) | NAB-PACLITAXEL (Phase II, Arm B)
Number analyzed (Participants) | 0 | 1 | 0
score on a scale |  | 0.47 [0.47 to 0.47] |

ADVERSE EVENTS:
Time Frame: 4 years
Description: RECIST criteria
Arm/Group | NAB-PACLITAXEL (Phase I) | PACLITAXEL (Phase II, Arm A) | NAB-PACLITAXEL (Phase II, Arm B)
All-Cause Mortality (participants affected / at risk) | 0/6 | 2/38 | 3/37
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/38 | 0/37
Other Adverse Events (participants affected / at risk) | 0/6 | 38/38 | 37/37
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NAB-PACLITAXEL (Phase I) (N=6) | PACLITAXEL (Phase II, Arm A) (N=38) | NAB-PACLITAXEL (Phase II, Arm B) (N=37)
acute respiratory failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
alanine aminotransferase increased (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 4 (4)
alopecia (Immune system disorders) | 0 (0) | 7 (7) | 9 (9)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 25 (25) | 26 (26)
anorexia (Gastrointestinal disorders) | 0 (0) | 10 (10) | 16 (16)
arthralgias (General disorders) | 0 (0) | 2 (2) | 2 (2)
aspartate aminotransferase increased (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 3 (3)
constipation (Gastrointestinal disorders) | 0 (0) | 5 (5) | 12 (12)
creatnine elevated (Blood and lymphatic system disorders) | 0 (0) | 4 (4) | 6 (6)
dercreased lymphocytes (Blood and lymphatic system disorders) | 0 (0) | 9 (9) | 13 (13)
decreased neutrophil count (Blood and lymphatic system disorders) | 0 (0) | 10 (10) | 25 (25)
decreased platelet count (Blood and lymphatic system disorders) | 0 (0) | 12 (12) | 19 (19)
dehydration (General disorders) | 0 (0) | 6 (6) | 5 (5)
decreased WBC (Blood and lymphatic system disorders) | 0 (0) | 8 (8) | 20 (20)
dermatitis (General disorders) | 0 (0) | 10 (10) | 10 (10)
diarrhea (Gastrointestinal disorders) | 0 (0) | 8 (8) | 6 (6)
dry mouth (General disorders) | 0 (0) | 1 (1) | 2 (2)
dysgeusia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 6 (6)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4)
albumin decreased (Blood and lymphatic system disorders) | 0 (0) | 8 (8) | 12 (12)
Alkaline phosphatase increased (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 4 (4)
hyponatremia (Blood and lymphatic system disorders) | 0 (0) | 7 (7) | 10 (10)
sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
thromboembolic event (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 3 (3)
Fever (General disorders) | 0 (0) | 4 (4) | 9 (9)
lymphocyte count decreased (Blood and lymphatic system disorders) | 0 (0) | 14 (14) | 22 (22)
chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 13 (13) | 16 (16)
pleural effusion (General disorders) | 0 (0) | 1 (1) | 2 (2)
sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 5 (5)
fatigue (General disorders) | 0 (0) | 19 (19) | 36 (36)
platelet count decreased (Blood and lymphatic system disorders) | 0 (0) | 12 (12) | 21 (21)
GERD (Gastrointestinal disorders) | 0 (0) | 6 (6) | 8 (8)
nausea (Metabolism and nutrition disorders) | 0 (0) | 12 (12) | 16 (16)
neutrophil count decreased (Blood and lymphatic system disorders) | 0 (0) | 9 (9) | 25 (25)
dizziness (Nervous system disorders) | 0 (0) | 4 (4) | 9 (9)
dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
dysphagia (General disorders) | 0 (0) | 16 (16) | 15 (15)
dyspnea (General disorders) | 0 (0) | 14 (14) | 19 (19)
edema feet (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1)
epistaxis (General disorders) | 0 (0) | 2 (2) | 3 (3)
esophageal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
esophagitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 16 (16) | 13 (13)
fecal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
gait disturbance (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
burning in mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
restless leg syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
anal fungal rash (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
seasonal allergies (General disorders) | 0 (0) | 0 (0) | 1 (1)
stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
post nasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
bilateral upper extremity lymphedema (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
abdominal cramping (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Heartburn (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
throat pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
vomiting (Gastrointestinal disorders) | 0 (0) | 9 (9) | 8 (8)
head congestion (General disorders) | 0 (0) | 0 (0) | 1 (1)
chest congestion (General disorders) | 0 (0) | 2 (2) | 1 (1)
difficulty swallowing (General disorders) | 0 (0) | 1 (1) | 0 (0)
BUN elevated (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
pleuritic pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
radiation fibrosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
right clavicular swelling (General disorders) | 0 (0) | 0 (0) | 1 (1)
Serum amylase increased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)

LIMITATIONS AND CAVEATS:
For Quality of life endpoints, we were limited by the log questionnaire completion rate. The number of patients completed quality of life questionnaire ranged from 1-8 patients in each are at month 3,6,9,12. Additionally, there was a high rate of missing data for FACT series questionnaire. As a result, we are reporting EQ-5D result at baseline and end of treatment.

The responsible party Dr. Hak Choy has been replaced with the Yuanyuan Zhang as Dr. Choy has left UTSouthwestern Medical Center.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-04): https://cdn.clinicaltrials.gov/large-docs/88/NCT01757288/Prot_SAP_000.pdf